CLINICAL TRIAL: NCT01423851
Title: A Phase 1/2, Open-label, Dose-Escalation Multi-center Study to Assess the Safety, Tolerability, PK and PD of Orally Administered NS-018 in Patients With Primary Myelofibrosis (MF), Post-polycythemia Vera MF, or Post-essential Thrombocythemia MF
Brief Title: Safety and Tolerability Study of Oral NS-018 in Patients With Primary Myelofibrosis (MF), Post-polycythemia Vera MF or Post-essential Thrombocythemia MF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NS-018-101
Record Dates: First submitted 2011-08-15; First posted 2011-08-26 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
Keywords: Keywords provided by NS Pharma, Inc.:; JAK2 kinase inhibitor; NS-018; Myeloproliferative Neoplasms; Primary Myelofibrosis; post-Polycythemia Vera Myelofibrosis; post-Essential Thrombocythemia Myelofibrosis; Additional relevant MeSH terms:; Bone Marrow Diseases; Hematologic Diseases; Polycythemia Vera; Thrombocythemia, Essential; PMF; post-PV MF; post-ET MF
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Polycythemia Vera; Thrombocythemia, Essential

STUDY DESIGN:
Intervention Model Description: Phase 1: 75, 125, 200, 300, 400 mg QD and 100, 200, 250, 300, 400 mg BID Phase 2: 300 mg QD
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention: Drug: NS-018 (Experimental): In Phase 1 part, subjects were treated with oral NS-018 at a dose of 75 - 400 mg once daily or 100 - 400 mg twice daily. In Phase 2 part, subjects were treated with oral NS-018 at a dose of 300 mg once daily.
  Interventions: Drug: NS-018

INTERVENTIONS:
Drug: NS-018 — Treatment will be administered continuously as oral daily therapy in cycles of 4 weeks in duration (28 day treatment cycles).

SUMMARY:
The purpose of this study is to determine the safety and tolerability of orally administered NS-018 in patients with Primary Myelofibrosis (PMF), Post-polycythemia Vera Myelofibrosis (post-PV MF), or Post-essential Thrombocythemia Myelofibrosis (post-ET MF)

DETAILED DESCRIPTION:
This is a Phase 1/2 study that is currently enrolling Janus kinase 2 (JAK2) failures into the Phase 2 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary myelofibrosis, post-PV MF, or post-ET MF that requires therapy
* MF patients must have received prior JAK2 inhibitor therapy, and been found to be intolerant, or refractory/relapsed from prior JAK2 inhibitor therapy, based on investigator assessment
* ≥18 years old
* ECOG Performance Status of ≤ 3
* Estimated life expectancy of ≥12 weeks
* Male or non-pregnant, non-lactating female patients
* Serum creatinine of ≤1.5 × the upper limit of normal (ULN)OR estimated creatinine clearance (CrCl) ≥ 40 ml/min/1.73 m2
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × the upper limit of normal (ULN) and total bilirubin ≤1.5 × ULN. If the total bilirubin is elevated between 1.5 x and 3 x ULN, patients with a direct bilirubin ≤ 1.5 X ULN are eligible during the Phase II portion.
* Absolute neutrophil count (ANC) >1000/μL and Platelet count > 25,000/μL
* QTcB ≤ 480 msec
* No MF-directed treatment for at least 2 weeks prior to initiation of NS-018, including any use of corticosteroids for Myelofibrosis symptom or blood count management. Low dose corticosteroids ≤ 10 mg/day prednisone or equivalent is allowed for non-myelofibrosis purposes.

Exclusion Criteria:

* Active, uncontrolled systemic infection
* Patients with any unresolved toxicity greater than Grade 1 from previous anticancer therapy
* Potentially curative therapy is available
* Currently taking medication that is substantially metabolized by cytochrome P450 (CYP) 1A2 or CYP3A4 or taking medication known to be strong inhibitors or inducers of CYP3A4
* Patients with a serious cardiac condition within the past 6 months
* Pregnant or lactating
* Radiation therapy for splenomegaly within 6 months prior to study entry
* Splenectomy (Phase 2 portion of the study only)
* Known HIV positive status
* Known active hepatitis, a history of viral hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-06; Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, M.D., Ph.D., Principal Investigator — MD Anderson Cancer Center, Houston, TX, 77030
Locations (9):
- United States (9):
  - Mayo Clinic Scottsdale Recruiting, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, San Diego, California
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York
  - MD Anderson Cancer Center, Department of Leukemia, Houston, Texas

REFERENCES:
- [Derived] Verstovsek S, Talpaz M, Ritchie E, Wadleigh M, Odenike O, Jamieson C, Stein B, Uno T, Mesa RA. A phase I, open-label, dose-escalation, multicenter study of the JAK2 inhibitor NS-018 in patients with myelofibrosis. Leukemia. 2017 Feb;31(2):393-402. doi: 10.1038/leu.2016.215. Epub 2016 Aug 1. PMID 27479177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were enrolled at 09 sites in the USA. The conduct of this study started on 02 June 2011 (the first patient screened) and the last patient last visit was on 22 April 2020.
  A total of 48 and 29 patients were enrolled during Phase 1 and Phase 2 of the study respectively.
  Participants could be reduced or escalated to the noted dose at physician discretion.
Pre-assignment Details: The screening period was from Day -14 to Day 0 for Phase I and Phase II. Informed consent form (ICF) was signed prior to screening procedures. All the study assessments were performed as per the schedule of assessment.
Groups:
- Part 1: 75 mg QD: Patients self-administered orally 75 mg of NS-018 once daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 125 mg QD: Patients self-administered orally 125 mg of NS-018 once daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 200 mg QD: Patients self-administered orally 200 mg of NS-018 once daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 300 mg QD; Part 2: 300 mg QD: Patients self-administered orally 300 mg of NS-018 once daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 400 mg QD: Patients self-administered orally 400 mg of NS-018 once daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 100 mg BID: Patients self-administered orally 100 mg of NS-018 twice daily (BID) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 200 mg BID: Patients self-administered orally 200 mg of NS-018 twice daily (BID) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 250 mg BID: Patients self-administered orally 250 mg of NS-018 twice daily (BID) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 300 mg BID: Patients self-administered orally 300 mg of NS-018 twice daily (BID) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
- Part 1: 400 mg BID: Patients self-administered orally 400 mg of NS-018 twice daily (BID) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
Period: Whole Study
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Started | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 8 | 8 | 8 | 29
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 8 | 8 | 8 | 29
Not completed — Disease progression | 2 | 1 | 1 | 4 | 1 | 3 | 1 | 4 | 0 | 2 | 10
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 3 | 4 | 12
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 3 | 2 | 3
Period: Dose Finding Period - Escalation
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Started | 0 | 1 | 4 | 4 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 4 | 4 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Period: Dose Finding Period - Reduction
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Started | 0 | 0 | 3 | 5 | 1 | 2 | 8 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 5 | 1 | 2 | 8 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 8 | 8 | 8 | 29 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: For Age continuous, Part 1 and Part 2 data are presented in different rows (48+29=77).
  Years
    Part 1: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 8 | 8 | 8 | 0 | 48
    Part 1 | 72.7 (1.5) | 70.3 (14.8) | 63.7 (12.9) | 67.3 (9.4) | 67.3 (3.8) | 65.0 (8.9) | 69.0 (3.6) | 63.0 (11.8) | 62.4 (11.9) | 69.3 (7.7) |  | 66.4 (9.6)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 29
    Part 2 |  |  |  |  |  |  |  |  |  |  | 67.2 (9.3) | 67.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 3 | 2 | 1 | 0 | 3 | 6 | 3 | 14 | 33
  Male | 3 | 2 | 3 | 3 | 1 | 2 | 3 | 5 | 2 | 5 | 15 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 3 | 3 | 2 | 6 | 2 | 3 | 2 | 8 | 8 | 8 | 26 | 71
  Black/African Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
  Asian/Oriental | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and Part 2: Number of Subjects With Adverse Events and Serious Adverse Event
Description: AEs (non-serious, serious) as variables of safety and tolerability of NS-018 were assesed. The number of patients were presented as Overall summary of AEs including treatment-emergent AEs (TEAEs); Treatment-emergent SAEs; Drug-related TEAEs; Treatment-emergent AEs leading to permanent discontinuation of study drug; Hospitalization or prolongation of existing hospitalization; Death.
Time Frame: From screening to until study discontinuation (approximate 8 years 10 months)
Population: The safety population included all patients who received at least 1 dose of study drug.
  NS-018-101 study was dose-finding study, Principal investigator (PI) could increase or decrease dose-level per protocol. Totals are based on number of patients and not on dose-level cohort. Patients can appear in more than one dose-level cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: 400 mg BID: Patients self-administered orally 400 mg of NS-018 once daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 3 | 4 | 10 | 15 | 4 | 5 | 13 | 8 | 12 | 8 | 29
Participants
  Not TEAE | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 4 | 2 | 6
  Any AE | 3 | 4 | 9 | 14 | 4 | 4 | 11 | 8 | 12 | 8 | 29
  Any Treatment Emergent AE | 3 | 4 | 9 | 14 | 4 | 4 | 11 | 8 | 12 | 8 | 29
  Drug Related TEAE | 1 | 1 | 8 | 11 | 4 | 2 | 4 | 5 | 10 | 7 | 24
  Any Serious TEAE | 2 | 2 | 2 | 6 | 1 | 1 | 4 | 3 | 4 | 3 | 13
  TEAE Leading to Discontinuation of study drug | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 3 | 4 | 2 | 5
  Hospitalization or Prolongation of Existing Hospitalization | 1 | 2 | 2 | 6 | 1 | 1 | 3 | 2 | 3 | 1 | 11
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Part 2: Number of Patient With Objective Response Using International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European Leukemia Net (ELN)
Description: Six response categories are listed: complete remission (CR) and partial remission signify treatment effects that are consistent with disease modification, whereas drug-induced improvements in MF-symptomatic burden were annotated as clinical improvement, anemia response, spleen response, orsymptoms response. Additional criteria are provided for progressive disease, stable disease, and relapse. The objective response was defined as the number of patients with confirmed complete remission (CR) + partial response (PR) + clinical improvement (CI) during the treatment period.
Time Frame: Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: The efficacy population included all patients who received at least one dose of study drug and had one baseline and at least one post-baseline efficacy assessment. Here, the overall number of subjects analyzed signifies only the subjects with available data that were analyzed evaluated on that specific cycle day.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 300 mg QD
Number analyzed (Participants) | 12
Participants | 1

3. Primary Outcome: Part 2: Change From Baseline in Spleen Size
Description: Change from baseline in spleen size was assessed by magnetic resonance imaging (MRI) (computed tomography [CT] scan for patients not able to tolerate MRI).
Time Frame: From Baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm3)
Arm/Group | Part 2: 300 mg QD
Number analyzed (Participants) | 16
cubic millimeter (mm3) | -335918.1 (558459.9)

4. Primary Outcome: Part 2: Change From Baseline in Bone Marrow Assessment
Description: Bone marrow was assessed by aspiration and biopsy for grade changes in osteomyelofibrosis. Fibrosis was graded according to European Consensus Myelofibrosis Grading Criteria, ranging from grade 0, which corresponds to normal bone marrow, to grade 3, in which coarse bundles of collagen fibrosis are identifiable with significant osteosclerosis.
Time Frame: From baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 300 mg QD
Number analyzed (Participants) | 3
Participants
  Increased by at least 1 grade level | 1
  Increased by at least 2 grade level | 0
  Decreased by at least 1 grade level | 2
  Decreased by at least 2 grade level | 0

5. Secondary Outcome: Part 1: Number of Patients With Objective Response Using International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT)
Description: Six response categories are listed: complete remission (CR) and partial remission signify treatment effects that are consistent with disease modification, whereas drug-induced improvements in MF-symptomatic burden were annotated as clinical improvement, anemia response, spleen response, orsymptoms response. Additional criteria are provided for progressive disease, stable disease, and relapse. The objective response was defined as the number of patients with confirmed "complete remission (CR) + partial response (PR) + clinical improvement (CI)" during the treatment period.
Time Frame: Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: The efficacy population included all patients who received at least one dose of study drug and had one baseline and at least one post-baseline efficacy assessment. NS-018-101 study was dose finding study, PI could increase or decrease dose-level per protocol. Patients can appear in more than one dose-level cohort.
  For 300 mg QD, data from 7 patients were available. 4 patients were enrolled originally and 2 patients were dose-reduced from 400 mg QD and 1 patient was dose-reduced from 250 mg BID.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID
Number analyzed (Participants) | 0 | 3 | 2 | 7 | 0 | 3 | 3 | 1 | 3 | 0
Participants | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0

6. Secondary Outcome: Part 1: Change From Baseline in Spleen Size
Description: Change from baseline in spleen size was assessed by palpation.
Time Frame: From Baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: The efficacy population included all patients who received at least one dose of study drug and had one baseline and at least one post-baseline efficacy assessment. NS-018-101 study was dose finding study, PI could increase or decrease dose-level per protocol. Patients can appear in more than one dose-level cohort.
  At 200 mg BID cohort, 3 patients were enrolled originally, 2 patients were dose-escalated from 100 mg BID cohort and 8 patients were dose-reduced from 300 mg BID or 400 mg BID cohort.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID
Number analyzed (Participants) | 0 | 3 | 2 | 6 | 0 | 3 | 13 | 1 | 3 | 0
cm |  | -0.67 (2.89) | -8.25 (3.18) | -3.17 (3.97) |  | -3.00 (3.00) | -4.33 (6.66) | -7.00 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | -2.00 (3.00) |

7. Secondary Outcome: Part 1: Change From Baseline in Bone Marrow Assessment
Description: as for outcome 4
Time Frame: From baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID
Number analyzed (Participants) | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 0 | 2 | 0
Participants
  Increased by at least 1 grade level |  | 0 |  | 1 |  | 1 |  |  | 2 |
  Increased by at least 2 grade level |  | 0 |  | 0 |  | 0 |  |  | 0 |
  Decreased by at least 1 grade level |  | 1 |  | 3 |  | 0 |  |  | 0 |
  Decreased by at least 2 grade level |  | 0 |  | 0 |  | 0 |  |  | 0 |

8. Secondary Outcome: Part 1: Change From Baseline in Quality of Life Assessments Using Myelofibrosis Symptom Assessment Form (MF-SAF)
Description: MF SAF is a 20-item instrument comprised of 4 subscales: 1) the Brief Fatigue Inventory [= average of 9 fatigue scores], 2) Splenomegaly associated symptoms [= average of 4 splenomegaly and associated scores], 3) Catabolic/proliferative Symptoms [= average of 3 catabolic/proliferative associated scores] and 4) Overall Quality of Life. The items were on a scale from 1 to 10 where 1= most favorable, and 10= least favorable.
Time Frame: From baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID
Number analyzed (Participants) | 0 | 3 | 2 | 7 | 0 | 3 | 2 | 1 | 3 | 0
score on a scale
  Brief Fatigue Inventory Score |  | 0.1 (0.4) | -1.3 (2.0) | 0.8 (1.3) |  | -1.9 (0.1) | 0.4 (0.2) | 0.7 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | -0.8 (1.1) |
  Splenomegaly-associated Symptom Score |  | 1.3 (1.3) | -0.5 (1.1) | 0.5 (0.8) |  | -0.3 (1.8) | -1.1 (1.2) | -4.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | -1.8 (1.5) |
  Catabolic/Proliferative Symptoms Score: number analyzed (Participants) | 0 | 2 | 2 | 7 | 0 | 3 | 2 | 1 | 3 | 0
  Catabolic/Proliferative Symptoms Score |  | 1.2 (0.2) | -0.7 (0.5) | -0.4 (2.4) |  | -0.4 (1.0) | 1.5 (1.6) | -8.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | -0.6 (1.0) |
  Overall Quality of Life Score: number analyzed (Participants) | 0 | 3 | 2 | 6 | 0 | 3 | 2 | 1 | 3 | 0
  Overall Quality of Life Score |  | 0.3 (0.6) | -1.0 (1.4) | 0.0 (3.6) |  | -1.7 (2.1) | -1.5 (2.1) | 0.0 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | -1.7 (1.5) |

9. Secondary Outcome: Part 2: Change From Baseline in Quality of Life Assessments Using Myeloproliferative Neoplasm Symptom Assessment Form (MPN SAF (MPN 10)
Description: Symptoms are evaluated by the MPN-SAF Total Symptom Score (TSS). The MPN-SAF TSS is assessed by the patients themselves and this includes fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers. Scoring is from 0 (absent/as good as it can be) to 10 (worst imaginable/as bad as it can be) for each item. The MPN-SAF TSS is the summation of all the individual scores (0-100 scale). Symptoms response requires >50% reduction in the MPN-SAF TSS.
Time Frame: From baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 2: 300 mg QD
Number analyzed (Participants) | 10
score on a scale | -0.7 (3.4)

10. Secondary Outcome: Part 1 and Part 2: Change in Baseline in Janus Kinase 2 (JAK2) V617F Allele Burden Levels
Description: The JAK2 V617F allele burden mean changes from baseline (%) are presented as pharmacodynamics parameters.
Time Frame: Part 1 and Part 2: From baseline to Cycle 7 Day 1 (duration of cycle was 4 weeks)
Population: The PD population included all patients who received at least one dose of study drug and had a baseline and at least one post-baseline PD assessment (for at least one PD parameter). Here, the overall number of subjects analyzed signifies only the subjects with available data that were analyzed evaluated on that specific cycle day.
Measure: Mean (Standard Deviation); unit: Percentage of JAK2 V617F Level
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 2 | 2 | 4 | 11
Percentage of JAK2 V617F Level |  | 4.360 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | -0.210 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | 7.410 (2.758) |  | -6.720 (10.479) | 8.255 (4.320) | -4.900 (9.065) | -9.033 (5.352) | -4.368 (14.602) | 1.782 (8.978)

11. Secondary Outcome: Part 2: Change From Baseline in Phosphorylated Signal Transducer and Activator of Transcription 3 (Phospho-STAT3)
Description: The Phospho-STAT3 mean changes from baseline (%) are presented as pharmacodynamics parameters.
  For phospho-STAT3 values (Phase 2 only), study samples were incubated (± IL-6) and labeled with CD markers. Surface markers included CD3+ (CD4+ [helper T cells] and CD8+ [cytotoxic T cells]) and CD14+ (monocytes) to which intracellular phospho STAT3 was targeted. The levels of phospho-STAT3 in CD14+, CD3+CD4+ and CD3+CD8+ cell subtypes were quantified. Phosphorylated-STAT3 levels were evaluated in the cell types before and after IL-6 incubation (stimulation) and reported both as mean fluorescence intensity (MFI) and the percentage of positive cells. For each sample time point, the MFI was normalized to a fold change.
  The fold change was calculated by MFI after IL-6 treatment/MFI before IL-6 treatment. The percent positive cells were normalized by subtracting the percent positive cells before IL-6 treatment from the percent positive cells after IL-6 treatment.
Time Frame: From Baseline to Pre-dose at Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 (duration of cycle was 4 weeks)
Population: The PD population included all patients who received at least one dose of study drug and had a baseline and at least one post-baseline PD assessment (for at least one PD parameter). Here, number analyzed reflects number of patients evaluated on that specific cycle day.
  Data from 17 out of 24 participants were available and contributed to the analysis. Samples from 7 patients were analyzed, but data were not available due to quantities not sufficient.
Measure: Mean (Standard Deviation); unit: Percentage of Phospho-STAT 3 Levels
Arm/Group | Part 2: 300 mg QD
Number analyzed (Participants) | 24
Percentage of Phospho-STAT 3 Levels
  Cycle 1 Day 1: Change percentage of Phospho-STAT3 Levels in CD14+ Positive cells: number analyzed (Participants) | 13
  Cycle 1 Day 1: Change percentage of Phospho-STAT3 Levels in CD14+ Positive cells | -9.406 (19.357)
  Cycle 1 Day 15: Change percentage of Phospho-STAT3 Levels in CD14+ Positive cells: number analyzed (Participants) | 11
  Cycle 1 Day 15: Change percentage of Phospho-STAT3 Levels in CD14+ Positive cells | -2.738 (16.191)
  Cycle 2 Day 1: Change percentage of Phospho-STAT3 Levels in CD14+ Positive cells: number analyzed (Participants) | 11
  Cycle 2 Day 1: Change percentage of Phospho-STAT3 Levels in CD14+ Positive cells | -0.422 (20.092)
  Cycle 1 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD4+ Positive cells: number analyzed (Participants) | 14
  Cycle 1 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD4+ Positive cells | -10.614 (11.178)
  Cycle 1 Day 15: Change percentage of Phospho-STAT3 Levels in CD3+ CD4+ Positive cells: number analyzed (Participants) | 12
  Cycle 1 Day 15: Change percentage of Phospho-STAT3 Levels in CD3+ CD4+ Positive cells | 6.217 (20.717)
  Cycle 2 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD4+ Positive cells: number analyzed (Participants) | 12
  Cycle 2 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD4+ Positive cells | -5.878 (16.304)
  Cycle 1 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD8+ Positive cells: number analyzed (Participants) | 14
  Cycle 1 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD8+ Positive cells | -3.707 (11.222)
  Cycle 1 Day 15: Change percentage of Phospho-STAT3 Levels in CD3+ CD8+ Positive cells: number analyzed (Participants) | 12
  Cycle 1 Day 15: Change percentage of Phospho-STAT3 Levels in CD3+ CD8+ Positive cells | 5.533 (14.513)
  Cycle 2 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD8+ Positive cells: number analyzed (Participants) | 12
  Cycle 2 Day 1: Change percentage of Phospho-STAT3 Levels in CD3+ CD8+ Positive cells | -1.644 (6.615)

12. Secondary Outcome: Part1 and Part 2: Observed Maximum Concentration (Cmax)
Description: To determine the Cmax as pharmacokinetic parameters of NS-018.
Time Frame: Pre-dose, 0.5 to 24 hours post-dose for Part 1: Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1 and for Part 2: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1 (duration of cycle was 4 weeks)
Population: The PK population include all patients who received at least one dose of study drug and have at least 50% of the planned samples above the limit of quantitation to provide evaluable PK profile, Here, number analyzed reflects number of patients evaluated on that specific cycle day.
  Part 2: 1 patient was completely excluded from PK Population due to critical samples missing, 1 patient was excluded from the analysis due to sample missing at timepoint, So the overall number of participants was 27.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 6 | 8 | 8 | 27
nanogram/milliliter (ng/mL)
  Cycle 1 Day 1 | 66.5600 (79.0171) | 404.5333 (26.4258) | 377.8000 (184.2086) | 726.0667 (232.0338) | 1643.0333 (789.0036) | 242.0333 (174.3374) | 351.0000 (257.1729) | 853.5833 (271.7900) | 1077.4750 (366.9158) | 1261.7000 (658.9141) | 957.9852 (306.7937)
  Cycle 1 Day 8 (Part 1 only): number analyzed (Participants) | 2 | 3 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 5 | 0
  Cycle 1 Day 8 (Part 1 only) | 30.6700 (13.3077) | 324.8667 (57.3280) | 539.6667 (160.0954) | 805.4333 (236.8877) | 1554.6667 (351.6765) | 412.8000 (232.9342) | 606.8333 (233.7812) | 806.8333 (464.3206) | 969.0167 (342.3090) | 1352.2200 (307.1358) |
  Cycle 1 Day 15 (Part 2 only): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 24
  Cycle 1 Day 15 (Part 2 only) |  |  |  |  |  |  |  |  |  |  | 732.5000 (313.5822)
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 5 | 2 | 23
  Cycle 2 Day 1 | 67.6467 (55.6250) | 450.6667 (187.4735) | 556.9000 (52.8463) | 1066.0000 (271.1854) | 1556.0000 (676.3941) | 408.6000 (127.0765) | 596.1333 (362.6751) | 830.7333 (166.0701) | 1272.5600 (420.7722) | 1040.6500 (321.5215) | 1035.3087 (445.9895)

13. Secondary Outcome: Part 1 and Part 2: Time to Maximum Plasma Concentration (Tmax)
Description: To determine the Tmax as pharmacokinetic parameters of NS-018.
Time Frame: Pre-dose, 0.5 to 24 hours post-dose for Part 1: Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1 and for Part 2: Cycle 1 Day 1, Cycle 2 Day 1 (duration of cycle was 4 weeks)
Population: as for outcome 12
Measure: Median (Full Range); unit: hours (h)
Groups:
- Part 1: 250 mg BID: Patients self-administered orally 250 mg of NS-018 twice daily (QD) in cycles of 28 days in duration (4 weeks) for Cycles 1, 2, 3, 4, 5, 6, 7 and until the patient experiences unacceptable toxicity that precludes any further treatment, disease progression, and/or as long as the patient is benefiting from treatment.
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 6 | 8 | 8 | 27
hours (h)
  Cycle 1 Day 1 | 1.00 [0.92 to 2.00] | 1.08 [1.00 to 2.00] | 2.00 [1.00 to 2.17] | 1.04 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 1.08] | 1.00 [1.00 to 1.00] | 1.46 [1.00 to 2.13] | 1.02 [1.00 to 23.58] | 2.00 [1.00 to 6.00] | 2.00 [0.92 to 3.00]
  Cycle 1 Day 8 (Part 1 only): number analyzed (Participants) | 2 | 3 | 3 | 6 | 3 | 3 | 3 | 6 | 6 | 5 | 0
  Cycle 1 Day 8 (Part 1 only) | 0.78 [0.50 to 1.05] | 1.00 [1.00 to 1.12] | 1.00 [1.00 to 2.00] | 1.54 [1.02 to 2.25] | 2.00 [1.00 to 2.05] | 1.00 [0.50 to 1.08] | 1.00 [0.50 to 1.02] | 1.98 [1.00 to 3.00] | 1.52 [0.83 to 4.42] | 2.03 [2.00 to 4.00] |
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 5 | 2 | 23
  Cycle 2 Day 1 | 1.00 [1.00 to 2.05] | 1.00 [1.00 to 2.03] | 1.00 [1.00 to 1.00] | 1.05 [0.83 to 2.00] | 1.00 [0.82 to 1.02] | 1.00 [0.53 to 1.00] | 1.00 [1.00 to 2.08] | 2.07 [1.00 to 4.00] | 2.08 [1.00 to 5.53] | 2.00 [1.00 to 3.00] | 1.08 [0.92 to 3.00]

14. Secondary Outcome: Part1 and Part 2: Area Under the Plasma Concentration-time Curve (AUC0-24)
Description: To determine the AUC0-24 as pharmacokinetic parameters of NS-018.
Time Frame: Pre-dose, 0.5 to 24 hours post-dose for Part 1: Cycle 1 Day 1, Cycle 2 Day 1 and for Part 2: Cycle 1 Day 1 (duration of cycle was 4 weeks)
Population: The PK Population includes all patients who received at least one dose of study drug and have at least 50% of the planned samples above the limit of quantitation to provide evaluable PK profile, regardless of whether derived from parent drug or metabolites.
  Part 2: One patient was completely excluded from the PK Population due to critical samples missing; Two patients were excluded from the analysis due to sample missing at time point. so the overall number of participants analyzed was 26.
Measure: Mean (Standard Deviation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 4 | 8 | 7 | 26
hour*nanogram/milliliter (h*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 2 | 3 | 4 | 8 | 7 | 26
  Cycle 1 Day 1 | 246.3454 (325.7347) | 1510.0507 (123.2939) | 1326.3929 (815.0175) | 2299.2216 (877.2554) | 5162.4119 (2485.9489) | 1022.0977 (521.6626) | 1241.5005 (461.6010) | 2117.1396 (449.2456) | 5666.7063 (5182.5571) | 7592.4070 (3031.4332) | 3672.2041 (1551.7435)
  Cycle 2 Day 1 (Part 1 only): number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 1 | 0
  Cycle 2 Day 1 (Part 1 only) | 253.6953 (306.7728) | 1905.2058 (938.2984) | 1816.8251 (559.9071) | 3175.6938 (794.6091) | 5443.2874 (986.8497) | 1561.1245 (621.5414) | 3470.6269 (2587.3663) | 5876.1106 (5133.4208) | 6132.2596 (3393.0644) | 3828.0995 (NA) — As only 1 participant was evaluable, hence SD is not calculable. |

15. Secondary Outcome: Part 1 and Part 2: Terminal Elimination Half-life (t½)
Description: To determine the t½ as pharmacokinetic parameters of NS-018.
Time Frame: as for outcome 13
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 6 | 7 | 7 | 27
hour (h)
  Cycle 1 Day 1 | 2.4878 (2.1008) | 5.1659 (0.5209) | 3.6685 (2.2953) | 4.4899 (1.5478) | 6.0302 (2.4730) | 9.7153 (5.2865) | 10.0780 (1.3932) | 5.9468 (3.8500) | 30.0521 (42.0129) | 13.4566 (7.3992) | 5.4384 (1.7469)
  Cycle 1 Day 8 (Part 1 only): number analyzed (Participants) | 2 | 3 | 3 | 6 | 3 | 3 | 3 | 5 | 6 | 4 | 0
  Cycle 1 Day 8 (Part 1 only) | 1.9170 (0.5066) | 2.4735 (0.3469) | 2.0217 (0.2653) | 2.6237 (0.5050) | 2.8480 (1.3889) | 2.3007 (0.0899) | 3.5204 (1.6584) | 2.6280 (0.8577) | 3.2062 (0.8054) | 2.8287 (1.2416) |
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 3 | 3 | 2 | 5 | 2 | 23
  Cycle 2 Day 1 | 3.7488 (2.9554) | 5.6743 (1.3845) | 5.4356 (0.7253) | 5.9316 (0.8500) | 8.5232 (5.0118) | 16.5535 (6.8417) | 8.7138 (6.8781) | 10.8357 (1.0282) | 13.7574 (8.1372) | 7.7683 (5.3755) | 2.8030 (1.2594)

16. Secondary Outcome: Part1 and Part 2: Accumulation Ratio (AR)
Description: To determine the AR as pharmacokinetic parameters of NS-018. AR was calculated as AR = (AUC0-24) Cycle 2 Day 1/ (AUC0-24) Cycle 1 Day 1.
Time Frame: Part 1 and Part 2: Cycle 2 Day 1 (duration of cycle was 4 weeks)
Population: The PK Population includes all patients who received at least one dose of study drug and have at least 50% of the planned samples above the limit of quantitation to provide evaluable PK profile (i.e. at least Cmax and AUC evaluable), regardless of whether derived from parent drug or metabolites.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 300 mg BID | Part 1: 250 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
Number analyzed (Participants) | 1 | 3 | 2 | 4 | 3 | 2 | 2 | 3 | 3 | 1 | 22
Ratio | 0.9778 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | 1.2517 (0.5579) | 1.1728 (0.0372) | 1.3581 (0.3108) | 1.2026 (0.4755) | 1.9941 (0.6140) | 3.3229 (0.3197) | 3.0501 (2.6306) | 1.5452 (0.4025) | 1.2514 (NA) — As only 1 participant was evaluable, hence SD is not calculable. | 1.0543 (0.2572)

ADVERSE EVENTS:
Time Frame: Part 1 and Part 2: From screening to until study discontinuation (approximate 8 years 10 months)
Description: Safety population: NS-018-101 study was dose finding study, PI could increase or decrease dose-level per protocol. Totals are based on number of patients and not on dose-level cohort. Patients can appear in more than one dose-level cohort.
Arm/Group | Part 1: 75 mg QD | Part 1: 125 mg QD | Part 1: 200 mg QD | Part 1: 300 mg QD | Part 1: 400 mg QD | Part 1: 100 mg BID | Part 1: 200 mg BID | Part 1: 250 mg BID | Part 1: 300 mg BID | Part 1: 400 mg BID | Part 2: 300 mg QD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/10 | 0/15 | 0/4 | 0/5 | 0/13 | 0/8 | 0/12 | 0/8 | 1/29
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 2/10 | 6/15 | 1/4 | 1/5 | 4/13 | 3/8 | 4/12 | 3/8 | 13/29
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 9/10 | 14/15 | 4/4 | 4/5 | 11/13 | 8/8 | 12/12 | 7/8 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 75 mg QD (N=3) | Part 1: 125 mg QD (N=4) | Part 1: 200 mg QD (N=10) | Part 1: 300 mg QD (N=15) | Part 1: 400 mg QD (N=4) | Part 1: 100 mg BID (N=5) | Part 1: 200 mg BID (N=13) | Part 1: 250 mg BID (N=8) | Part 1: 300 mg BID (N=12) | Part 1: 400 mg BID (N=8) | Part 2: 300 mg QD (N=29)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulval cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 75 mg QD (N=3) | Part 1: 125 mg QD (N=4) | Part 1: 200 mg QD (N=10) | Part 1: 300 mg QD (N=15) | Part 1: 400 mg QD (N=4) | Part 1: 100 mg BID (N=5) | Part 1: 200 mg BID (N=13) | Part 1: 250 mg BID (N=8) | Part 1: 300 mg BID (N=12) | Part 1: 400 mg BID (N=8) | Part 2: 300 mg QD (N=29)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 6 | 1 | 1 | 3 | 1 | 4 | 3 | 11
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 1 | 0 | 2 | 3 | 7 | 1 | 10
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 3 | 2 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 0 | 0 | 1 | 2 | 2 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 8
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 5 | 1 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal sphincter atony (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Blood potassium increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Physical examination abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart rate abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B1 decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 5 | 1 | 1 | 4 | 4 | 3 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 5 | 0 | 2 | 2 | 1 | 4 | 2 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic girdle pain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 6 | 1 | 2 | 3 | 2 | 4 | 2 | 11
Oedema peripheral (General disorders) | 1 | 0 | 2 | 5 | 0 | 2 | 1 | 2 | 1 | 0 | 10
Pyrexia (General disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 0 | 3
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Oedema (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Nodule (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 2 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 2 | 0 | 1 | 0 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 5 | 2 | 2 | 3 | 3 | 6 | 2 | 8
Headache (Nervous system disorders) | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 1 | 5 | 1 | 11
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 3
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 3 | 1 | 2 | 5 | 2 | 6 | 3 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 3 | 1 | 4
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 4 | 2 | 1 | 1 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 5 | 0 | 1 | 2 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Genital abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infected seroma (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 4
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Claustrophobia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep terror (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tobacco withdrawal symptoms (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 3
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This confidential document is the property of NS Pharma, Inc. No unpublished information contained herein may be disclosed without prior written approval from NS Pharma, Inc. Access to this document must be restricted to relevant parties.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT01423851/Prot_SAP_000.pdf